CLINICAL TRIAL: NCT01299935
Title: Stress Reduction and Cardiovascular Disease Morbidity and Mortality
Brief Title: A Randomized Controlled Trial of Stress Reduction on Cardiovascular Morbidity and Mortality in African Americans
Acronym: Milw
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director, Center for Natural Medicine and Prevention, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01HL048107 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Coronary Heart Disease; Cardiovascular Disease
Keywords: stress reduction; Transcendental Meditation technique; secondary prevention of coronary heart disease
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases | interventions — Meditation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress reduction (Experimental): Stress reduction program utilizing the Transcendental Meditation (TM) technique
  Interventions: Behavioral: Transcendental Meditation
- health education (Active Comparator): health education is taught in a clinical setting using standard AHA recommendations for proper diet, exercise and control of substance usage but without a stress management component.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Transcendental Meditation — The Transcendental Meditation program is the principal mind-body approach of Maharishi Ayurveda, originating from the ancient Vedic tradition and introduced 50 years ago by Vedic scholar and teacher Maharishi Mahesh Yogi. The Transcendental Meditation technique is described as a simple and natural procedure that is practiced 20 minutes twice a day while sitting comfortably with the eyes closed. Practice of the Transcendental Meditation technique does not require any changes in personal beliefs, philosophy or lifestyle. During the practice a unique state of restful alertness is gained. Acute and chronic physiological effects have been documented. The course is taught by instructors certified by Maharishi Foundation - USA.
  Other Names: Transcendental Meditation technique, TM technique
  Arms: Stress reduction
Behavioral: Health Education — health education is taught in a clinical setting using standard AHA recommendations for proper diet, exercise and control of substance usage but without a stress management component.
  Other Names: lifestyle modification
  Arms: health education

SUMMARY:
This randomized controlled clinical trial tests the hypothesis that a selected stress reduction approach, the Transcendental Meditation program will reduce all-cause mortality, myocardial infarction and stroke in African American patients with coronary heart disease. Secondary hypotheses include effects on other cardiovascular clinical events, blood pressure and psychosocial stress.

DETAILED DESCRIPTION:
The overall objective of this randomized controlled trial is to conduct a long-term evaluation of the effects of the Transcendental Meditation (TM) program compared to health education (HE) on secondary prevention of clinical events in African American men and women with coronary artery disease (CAD). Patients (N=201; mean age 59 yrs) were enrolled with documented CAD (i.e., coronary angiogram showing at least one artery with > 50% stenosis). Patients were pretested at baseline and every 6-12 months for the duration of the study for incidence of clinical events, BP, BMI, medication usage, lifestyle behaviors, psychosocial stress factors and intervention compliance. Subjects were followed for a maximum of 9.2 years (mean 5.4 years). The investigators hypothesize that a selected stress reduction intervention, the TM program compared with a health education control may significantly reduce risk for death, myocardial infarction (MI) and stroke in African American men and women with CHD. If successful, the Transcendental Meditation program may be clinically useful in the secondary prevention of cardiovascular disease in a high-risk population.

ELIGIBILITY:
Inclusion Criteria:

African American men and women with documented coronary heart disease defined a coronary angiogram demonstrating the presence of one more coronary arteries with > or = 50% stenosis.

Exclusion Criteria:

acute MI, stroke or coronary revascularization within the previous three months; symptomatic heart failure with EF < 20%; dementia or other cognitive impairment determined clinically; and non-cardiac life threatening illness.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 1998-01; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
composite of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke | every six months for an average of 5.4 years

SECONDARY OUTCOMES:
composite of cardiovascular mortality, nonfatal MI, nonfatal stroke, coronary revascularization, and hospitalization for heart failure, unstable angina or ischemic heart disease - non-MI. | every six months for average of 5.4 years
psychosocial distress factors | annually for an average of 5.4 years
  psychometric factors included depression, hostility and anger using standardized psychometric instruments - Center for Epidemiological Depression Scale (CES-D), Cook-Medley Hostility Inventory (Ho), Anger Expression Scale (AX)
blood pressure | every six months for an average of 5.4 years
  BP was assessed by standard clinical trial technique using multiple seated measurements in the research clinic
behavioral and lifestyle factors | annually for an average of 5.4 years
  smoking, alcohol use, physical activity and dietary patterns were assessed by standard questionnaire. Body mass index was measured by balance and scale.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Schneider RH, Grim CE, Rainforth MV, Kotchen T, Nidich SI, Gaylord-King C, Salerno JW, Kotchen JM, Alexander CN. Stress reduction in the secondary prevention of cardiovascular disease: randomized, controlled trial of transcendental meditation and health education in Blacks. Circ Cardiovasc Qual Outcomes. 2012 Nov;5(6):750-8. doi: 10.1161/CIRCOUTCOMES.112.967406. Epub 2012 Nov 13. PMID 23149426